CLINICAL TRIAL: NCT04673903
Title: The Effect of the Copenhagen Adduction Exercise on Groin Injuries Rate Among Soccer Players. A Cluster Randomized Controlled Trial.
Brief Title: The Effect of the Copenhagen Adduction Exercise on Groin Injuries Rate Among Soccer Players.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Wesam Saleh A. Al Attar, PT, MSc, PhD, Professor, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HAPO-02-K-012-2020-11-481
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Groin Injuries
Keywords: Copenhagen Adduction Exercise; Groin injuries; Soccer

STUDY DESIGN:
Intervention Model Description: The intervention group will be instructed to include the Copenhagen adduction exercise into their warm up before training session (3 times per week) during one season (6 months).The control group will practice their usual warm up.
  Usual warm up is defined as any basic exercises performed before a performance or practice to prepare the muscles for vigorous actions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will be instructed to include the Copenhagen adduction exercise into their warm up before training session (3 times per week) during one season (6 months).
  The Copenhagen adduction exercise is a body-weight exercise which mainly works the groin and hip adductor. It has a large eccentric component, meaning the muscles are working whilst lengthening.
  Interventions: Other: Copenhagen adduction exercise
- Control group (Active Comparator): The control group will practice their usual warm up. Usual warm up is defined as any basic exercises performed before a performance or practice to prepare the muscles for vigorous actions.
  Interventions: Other: Usual warm up

INTERVENTIONS:
Other: Copenhagen adduction exercise — The Copenhagen Adduction exercise is a simple isolated eccentric partner exercise and doesn't require special equipment and can be performed as a warm up activity on the pitch.
  Arms: Intervention group
Other: Usual warm up — Usual warm up is defined as any basic exercises performed before a performance or practice to prepare the muscles for vigorous actions.
  Arms: Control group

SUMMARY:
The effect of the Copenhagen Adduction Exercise on groin injuries rate among soccer players The Copenhagen adduction exercise is a body-weight exercise which mainly works the groin and hip Adductors. It has a large eccentric component, meaning the muscles are working whilst lengthening.

The purpose of this study is to investigate the effect of the Copenhagen adduction exercise on groin injuries among soccer players.

It hypothesized that Copenhagen adduction exercise has a beneficial effect in terms of groin injury prevention.

DETAILED DESCRIPTION:
Study type Interventional Description of intervention(s) / exposure The intervention group will be instructed to include the Copenhagen adduction exercise into their warm up before training session (3 times per week) during one season (6 months).

Group sessions will be administered by an exercise physiologist and/ or athletic trainer and/ or soccer coaches and/ or strength and conditioning specialists and/ or physiotherapist.

Session attendance checklists will be used to assess or monitor adherence to the intervention.

The Copenhagen adduction exercise is a body-weight exercise which mainly works the groin and hip adductor. It has a large eccentric component, meaning the muscles are working whilst lengthening.

The Copenhagen Adduction exercise is a simple isolated eccentric partner exercise and doesn't require special equipment and can be performed as a warm up activity on the pitch.

The Copenhagen Adduction exercise requires a partner who will hold the player's upper leg in an extended position nearly at the hip level of the partner, with one hand supporting the knee and the other upholding the ankle. Meanwhile, the player will lie on one side and support the body with the forearm on the ground and the top arm being placed along the body. Then, the player will elevate the trunk from the floor and raise the lower leg in a straight line. The player will repeat this for 3 seconds until the feet touch each other. This will be followed by slightly lowering the body just to the ground for 3 seconds until it touches the level of the foot.

It must be performed on both limbs. It is crucial to note that the most accurate performance of the exercise must avoid trunk bending. In terms of the training form, the frequency is three-two sessions per week while the repetition varies according to the different levels of the players ranging from 3-12 times in one-two sets.

Prevention Comparator / control treatment The control group will practice their usual warm up. Usual warm up is defined as any basic exercises performed before a performance or practice to prepare the muscles for vigorous actions.

ELIGIBILITY:
Inclusion Criteria:

Soccer teams Amateur. Male . Training at least three times per week.

Exclusion Criteria:

History of lower extremity injury requiring medical attention in the past 6 months, or systemic diseases, cardiovascular disease, neurological disorders or bone fractures or surgery in the previous year.

Players who joined a participating team after the start of the trial will be excluded.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-01-16 (Estimated); Primary Completion 2021-06-16 (Estimated); Study Completion 2021-07-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of initial injuries | At the end of the intervention season (6 months)
  Injury is defined according to a consensus statement on injury definitions and data collection procedures in soccer studies; an injury will be recorded if it caused the player to be unable to completely participate in the following match or training session.Injury rates will be summarised as number of injuries per 1000 player-hours for both matches and training. Exposure time in hours will be calculated for each team over a 6-month period.
  Data will be collected from Sports Injury Tracker injury reporting form. Coaches in both the experimental and control groups will be reporting injuries during training and matches by filling in forms once per week and submitting the information using the Sports Injury Tracker injury reporting form (Sports Medicine Australia).
  Injury rates will be summarised as number of injuries per 1000 player-hours for both matches and training. Exposure time in hours will be calculated for each team over a 6-month period.
The incidence of recurrent injuries | At the end of the intervention season (6 months)
  Recurrent injury is defined as a repeat episode of a fully recovered injury. Injury is defined according to a consensus statement on injury definitions and data collection procedures in soccer studies; an injury will be recorded if it caused the player to be unable to completely participate in the following match or training session.
  Data will be collected from Sports Injury Tracker injury reporting form.

SECONDARY OUTCOMES:
Injury severity | At time of any injury occurring throughout intervention soccer season (6 months)
  Defined as time loss in days (days unable to train): minor (1 to 7 days lost), moderate (8 to 21 days lost), or severe (>21 days lost). Injury severity data will be collected from Sports Injury Tracker injury reporting form.
Compliance with the intervention | At the end of the intervention season (6 months)
  The rate of compliance using attendance log.

CONTACTS AND LOCATIONS:
Locations (1):
- Umm Al Qura University, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Start: Immediately following publication for 5 years.
Access Criteria: Access subject to approvals by Principal Investigator. The Principal Investigator can be contacted by email wsattar@uqu.edu.sa

REFERENCES:
- [Background] Ishoi L, Sorensen CN, Kaae NM, Jorgensen LB, Holmich P, Serner A. Large eccentric strength increase using the Copenhagen Adduction exercise in football: A randomized controlled trial. Scand J Med Sci Sports. 2016 Nov;26(11):1334-1342. doi: 10.1111/sms.12585. Epub 2015 Nov 21. PMID 26589483
- [Background] Haroy J, Clarsen B, Wiger EG, Oyen MG, Serner A, Thorborg K, Holmich P, Andersen TE, Bahr R. The Adductor Strengthening Programme prevents groin problems among male football players: a cluster-randomised controlled trial. Br J Sports Med. 2019 Feb;53(3):150-157. doi: 10.1136/bjsports-2017-098937. Epub 2018 Jun 10. PMID 29891614
- [Background] Holmich P, Uhrskou P, Ulnits L, Kanstrup IL, Nielsen MB, Bjerg AM, Krogsgaard K. Effectiveness of active physical training as treatment for long-standing adductor-related groin pain in athletes: randomised trial. Lancet. 1999 Feb 6;353(9151):439-43. doi: 10.1016/S0140-6736(98)03340-6. PMID 9989713
- [Background] Holmich P. Groin injuries in athletes--development of clinical entities, treatment, and prevention. Dan Med J. 2015 Dec;62(12):B5184. PMID 26621401
- [Background] Haroy J, Thorborg K, Serner A, Bjorkheim A, Rolstad LE, Holmich P, Bahr R, Andersen TE. Including the Copenhagen Adduction Exercise in the FIFA 11+ Provides Missing Eccentric Hip Adduction Strength Effect in Male Soccer Players: A Randomized Controlled Trial. Am J Sports Med. 2017 Nov;45(13):3052-3059. doi: 10.1177/0363546517720194. Epub 2017 Aug 14. PMID 28806100